CLINICAL TRIAL: NCT03053960
Title: Predictability of Carcinomatous Invasion of the Maxilla or Mandible: An Assessment of Radiologic Modalities With Histologic Correlation
Brief Title: Helical CT, PET/CT, MRI, and CBCT Alone or in Combination in Predicting Jaw Invasion in Patients With Oral Cancer
Status: Terminated | Type: Observational
Why Stopped: Terminated by IRB
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Other Study IDs: 15D.468; JT 6307 (Other: JeffTrial Number)
Record Dates: First submitted 2017-01-31; First posted 2017-02-15 (Actual); Results first posted 2019-12-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Oral Cavity Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Tomography, X-Ray Computed; Positron Emission Tomography Computed Tomography; Cone-Beam Computed Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnostic (helical CT, PET/CT, MRI, CBCT): Patients undergo helical (Computed Tomography) CT,(Positron Emission Tomography and Computed Tomography) PET/CT, (Magnetic Resonance Imaging) MRI, and (Cone-Beam Computed Tomography) CBCT scans. Patients also undergo therapeutic conventional surgical resection of tumor.
  Interventions: Device: Computed Tomography; Device: Positron Emission Tomography and Computed Tomography Scan; Device: Cone-Beam Computed Tomography; Device: Magnetic Resonance Imaging; Procedure: Therapeutic Conventional Surgery; Procedure: Histopathologic Examination

INTERVENTIONS:
Device: Computed Tomography — Undergo helical CT scan
  Other Names: CAT Scan; Computerized Axial Tomography; CAT
Device: Positron Emission Tomography and Computed Tomography Scan — Undergo PET/CT scan
  Other Names: PET-CT Scan; PET/CT SCAN
Device: Cone-Beam Computed Tomography — Undergo CBCT scan
Device: Magnetic Resonance Imaging — Undergo MRI scan
  Other Names: MRI; MRI Scan
Procedure: Therapeutic Conventional Surgery — Undergo resection of tumor
Procedure: Histopathologic Examination — Correlative studies
  Other Names: Histopathologic Study

SUMMARY:
This clinical trial studies how well helical computed tomography (CT), positron emission tomography (PET)/CT, magnetic resonance imaging (MRI), and cone beam computed tomography (CBCT) work alone or in combination in predicting whether tumor cells have spread to the jaw bone (jaw invasion) in patients with oral cancer. Imaging, such as helical CT, PET/CT, MRI, and CBCT, may help find out how far cancer has spread. Accurate prediction of the presence or absence of jaw invasion may help create a better surgical treatment plan for patients with oral cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine which imaging modality or combination of imaging methods, in conjunction with clinical and histological examination, will most accurately predict the presence or absence of invasion of the mandible or maxilla by intraoral squamous cell carcinoma (SCC).

SECONDARY OBJECTIVES:

I. To compare the histopathologic findings to the radiologic findings.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of squamous cell carcinoma of the oral cavity
* Able to read and sign and informed consent

Exclusion Criteria:

* Prior mandibular surgery
* Primary intraosseous carcinoma
* Prior history of radiation to the mandible
* Obvious finding of clinical invasion of the mandible

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data from all of the subjects that are enrolled and have consented to be a part of the study will be analyzed
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Gold, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (Helical CT, PET/CT, MRI, CBCT)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Helical CT, PET/CT, MRI, CBCT)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Accurate Predication of the Presence or Absence of Bone Invasion by Oral Squamous Cell Carcinoma by Helical CT, PET/CT, MRI and CBCT
Description: Sensitivity and specificity of the clinical exam, CBCT, helical CT, PET/CT, MRI and any other imaging modality used in detection of bone invasion will be calculated, as compared to the histological examination of the specimens. The positive and negative predictive value will be calculated for each modality using the true positive and negatives as well as false positive and negative values
Time Frame: Up to 2 years
Population: The study was terminated by the IRB. Sincere efforts were made to gather and report the data, however, no data is available for the study.
Arm/Group | Diagnostic (Helical CT, PET/CT, MRI, CBCT)
Number analyzed (Participants) | 0

2. Secondary Outcome: Incidence of Sparing Resection
Time Frame: Up to 2 years
Population: as for outcome 1
Arm/Group | Diagnostic (Helical CT, PET/CT, MRI, CBCT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: baseline to 30 days after completion of study treatment
Arm/Group | Diagnostic (Helical CT, PET/CT, MRI, CBCT)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT03053960/Prot_SAP_000.pdf